CLINICAL TRIAL: NCT01062789
Title: Use of an Optical Breath-hold Control (OBC) System for Image-guided Interventional Radiology Procedures: A Feasibility Study
Brief Title: Optical Breath-hold Control System for Image-guided Procedures
Acronym: OBC
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Closed due to funding and never enrolled a subject
Sponsor: Mayo Clinic (Other)
Responsible Party: Stephanie K. Carlson, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-004069
Record Dates: First submitted 2010-01-28; First posted 2010-02-04 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Respiration
Keywords: lung biopsy; computed tomograph; respiratory motion; Controlling respiratory motion in CT guided lung biopsies; biopsy
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Use of an optical breath-hold control device (Other): This is a feasibility study that will use this new device in place of a different bellows-based breath-hold control device for a series patients undergoing CT-guided lung biopsy. The new belt will be used in all patients in our study.
  Interventions: Device: Optical breath-hold control system (OBC)

INTERVENTIONS:
Device: Optical breath-hold control system (OBC) — The OBC system was designed to replace the IBC rubber bellows respiration sensor system that we are currently using for CT-guided lung biopsies. Unlike the IBC, the OBC is 1) unaffected by temperature changes, 2) has a linear sensitivity (for easier use and better accuracy), 3) has no pneumatic purge time when setting reference breath-hold level (reducing the chance of an inappropriate reference), 4) has no pneumatic cable that can occasionally interfere and get pinched during procedures, 5) is ambulatory (so patients can more easily familiarize themselves with the device before the procedure), 6) is capable of indicating proper fitting tension, 7) allows for easier binding (wireless pairing with other system components), and 8) is significantly less expensive (and possibly disposable).

SUMMARY:
The objective or our study is to test the feasibility of a new optical-based breath-hold control (OBC) system for monitoring breath-hold levels and providing patient feedback during CT-guided biopsies of the lung and upper abdomen where respiratory motion is a problem.

DETAILED DESCRIPTION:
1. Specific Aim #1: To further test the feasibility of the new OBC system for guiding accurate and reproducible breath-hold levels that correlate with internal target position in human volunteers. Hypothesis: The OBC system is as good as or better than the currently used IBC system with regard to accuracy and reproducibility of a reference breath-hold level.
2. Specific Aim #2: To compare the use of 2 optical-based belts (wrapped around the chest and abdomen) versus 1 optical-based belt (wrapped around the chest or abdomen, depending on which region expands the most during respiration) with regard to accuracy and reproducibility of a pre-determined reference breath-hold level in a subset of patients (prone and/or obese). Hypothesis: The use of 2 optical-based belts allows increased accuracy and reproducibility of a pre-determined reference breath-hold level compared with the use of only one belt in this subset of patients.
3. Specific Aim #3: To test the clinical feasibility of the new OBC system in patients undergoing CT-guided biopsy of the lung or upper abdomen where respiratory motion is a problem. Hypothesis: The OBC system is as good as or better than the currently used IBC system with regard to the accuracy and reproducibility of the reference breath-hold and ease of use.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for a CT-guided lung or upper abdomen biopsy (including lesions in the liver, pancreas, stomach, kidneys, adrenals, spleen, or in the peritoneum at or above the level of the kidneys) on the SMH-CT-3M scanner when either Dr. Carlson or Dr. Bender are scheduled.
* Lesions will need to measure 3 cm or less in maximum dimension and cannot be affixed to the chest or abdominal wall.

Exclusion Criteria:

* Inability to cooperate with breath-holding (including cognitive impairment, poor pulmonary function that inhibits patients from being able to hold their breath for at least 10 seconds)
* Patients with bleeding diatheses (platelets < 50,000, International Normalized Ratio > 1.5, or activated partial thromboplastin time > twice normal)
* Lesions that abut the pleura or abdominal wall for a distance greater than 3 cm (these lesions were assumed to be fixed in position and less likely to be affected by respiratory motion).
* Patients with implanted medical devices (pacemakers) (this exclusion is based on the Division of Engineering Safety Review-enclosed in application)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Ability to monitor patient respiration (return of target to same anatomical position) | Measured daily for each individual procedure

SECONDARY OUTCOMES:
Needle Placement Time | Measured daily for each individual procedure

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie K Carlson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States